CLINICAL TRIAL: NCT04455802
Title: Prospective Randomized Blinded Trial to Shorten Pharmacologic Treatment of Newborns With Neonatal Opioid Withdrawal Syndrome (NOWS)
Brief Title: Randomized Control Trial of Buprenorphine vs. Morphine for the Treatment of Neonatal Opioid Withdrawal Syndrome (NOWS)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: termination of funding
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, James Padbury, Principal Investigator, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WIH 19-0042; 1P20GM125507-01 (NIH)
Record Dates: First submitted 2020-06-08; First posted 2020-07-02 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Neonatal Opioid Withdrawal Syndrome
Keywords: Neonatal Opioid Withdrawal Syndrome; Neonatal Abstinence Syndrome
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Buprenorphine; Morphine

STUDY DESIGN:
Intervention Model Description: Infants will be randomly assigned to treatment arms of either morphine or buprenorphine
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be a randomized, double-blind, double-dummy, intention-to-treat clinical trial. All clinical providers, research personnel and participants will be blinded to group assignment. Pharmacy personnel will be the only un-blinded individuals. The placebo medication will be identical in appearance and volume to a dose of the medication at the respective dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Morphine (Active Comparator): Infants randomized to the morphine arm will start at a dose of 0.06 mg/kg/dose every 4 hours. A buprenorphine placebo will also be given at the same frequency as a faux drug.
  Interventions: Drug: Buprenorphine or Placebo; Drug: Morphine or Placebo
- Buprenorphine (Experimental): Infants randomized to the buprenorphine arm will be started on a dose of 10 mg/kg/dose every 8 hours. A morphine placebo will also be given at the same frequency as a faux drug.
  Patients can only be randomized to only one arm.
  Interventions: Drug: Buprenorphine or Placebo; Drug: Morphine or Placebo

INTERVENTIONS:
Drug: Buprenorphine or Placebo — The double blind, double dummy design necessitates that both drugs be on an identical schedule. The 4-hour dosing allows for this pairing. If a patient is randomized to the buprenorphine arm, medication administration will follow an every 8-hour dosing but medication will be substituted with placebo during the intermediary time point.
Drug: Morphine or Placebo — If a patient is randomized to the morphine arm, morphine will be given every 4 hours. Placebo will also be given at the same frequency as a faux drug.

SUMMARY:
This randomized control trial will compare buprenorphine and morphine, two currently used medications for the treatment of neonatal opioid withdrawal syndrome (NOWS), in newborns to determine which medication will reduce the number of days of pharmacological treatment.

DETAILED DESCRIPTION:
This randomized control trial will compare buprenorphine to morphine, two currently used medications for the treatment of NOWS, to determine whether the use of buprenorphine for NOWS treatment will reduce the number of days of pharmacological treatment. After an infant is born they will be monitored for signs of NOWS. Once an infant reaches treatment thresholds, they will be randomized using a double dummy design to either the buprenorphine or morphine treatment arm. After randomization infants will receive a syringe with either morphine or placebo every 4 hours and every 8 hours infant will receive 1 sublingual application of buprenorphine or placebo. To maintain the blind infants enrolled in the study will receive both interventions. During the study medication doses will be weaned by 10% of the stabilization dose. Study intervention will continue until 20 percent of the maximal dose has been reached. Use of a second line drug will be permissible after randomization and after an infant has had 2 consecutive escalations. Second line drug will be phenobarbital, in addition to the study drug. Infants in both groups will be evaluated and scored for NOWS symptoms to determine if weaning study medication is permissible each day. NOWS scores that do not reach the threshold for escalation will wean in accordance with standard clinical practice. If NOWS symptoms increase during treatment, infants will have the dose of the study drug increased by 10% to the previous day's dose. When stable for 24 hours, the weaning process will continue. The NICU Network Neurobehavioral Scale (NNNS) will be administered prior to starting study medication and once off study medication but prior to discharge to examine proportion of infants in each medication arm for the abnormal NNNS profiles which has been associated with atypical early childhood outcomes including behavior problems and low IQ scores. Development at 18 months of age will also be assessed to examine any differences in both arms of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Infant gestational age greater than or equal 36 weeks
2. Mother receiving either methadone from a drug treatment program, buprenorphine from a licensed physician, or an opioid prescription for a documented medical need
3. Mother had at least 2 prenatal appointments.
4. Infant toleration of oral medication administration
5. Infant is considered medically stable by the attending physician
6. Singleton Pregnancy
7. English Speaking

Exclusion Criteria:

1. Within 30 days of birth the mother has actively used illicit drugs (excluding THC) or obtaining oral opioids, methadone, or buprenorphine from a non-licensed physician or drug treatment program
2. The mother has had less than 2 prenatal care visits
3. The mother reports excessive alcohol use during pregnancy
4. Mother is less than 18 years of age or is not capable of signing consent
5. The infant has a gestational age less than or equal to 35 weeks and 6 days
6. The infant has dysmorphic features including evidence of aneuploidy
7. The infant is not able to tolerate oral medication administration
8. Multiple gestation pregnancy
9. Hypoxic-ischemic encephalopathy
10. Seizures from etiologies other than NOWS
11. Non-English Speaking
12. Infant started on NOWS standard care medication prior to study consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Total amount of opioid medication for treatment of NOWS | Duration of pharmacological treatment with opioid medication while admitted to the hospital up to 30 days
  Total amount of opioid medication given to infant for the duration of their hospitalization

SECONDARY OUTCOMES:
Length of total stay | During hospitalization for NOWS up to 30 days
  Length of hospital stay due to NOWS
Length of stay secondary to NOWS | During hospitalization for NOWS up to 30 days
  Total length of hospital stay secondary to NOWS
Neurobehavioral Profile | At birth before randomization to NOWS treatment arm around 18-24 hours of life and prior to hospital discharge up to 30 days of life
  Neurobehavior will be assessed with Neonatal Intensive Care Unit (NICU) Network Neurobehavioral Scale (NNNS). The NNNS is a comprehensive evaluation of neurologic and behavioral functioning as well as signs of stress. Profile 5 is the most atypical, and is characterized by exaggerated scores for arousal, excitability, hypertonicity, quality of movement, and stress abstinence. The atypical profile as been associated with atypical early childhood outcomes, including more behavior problems and lower IQ scores. Researchers will compare the proportion of atypical neurobehavioral profiles for infants in each intervention arm.
Cognitive, Language, and Motor Development From 18 Month Old Bayley Neurodevelopmental Assessment | 18 months old
  The Bayley Scales of Infant and Toddler Development (BSID-III) assesses the development of infants and children (1-42 months) through a series of developmental play tasks, identifying children with developmental delay. Raw scores of completed items are summarized within three distinct scale scores (Cognitive Scale, Language Scale, Motor Scale). Scale scores are each converted to composite scores to determine the child's performance compared with scores of age-matched children of typical development (percentile rank). A higher composite score indicates more ideal developmental outcome (range 40-160). At 18 month follow-up visit, participants were assessed using the BSID-III for composite score outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Czynski, DO, Principal Investigator — Women and Infants Hospital
Locations (1):
- Women and Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lester BM, Tronick EZ, Brazelton TB. The Neonatal Intensive Care Unit Network Neurobehavioral Scale procedures. Pediatrics. 2004 Mar;113(3 Pt 2):641-67. PMID 14993524
- [Background] Davis JM, Shenberger J, Terrin N, Breeze JL, Hudak M, Wachman EM, Marro P, Oliveira EL, Harvey-Wilkes K, Czynski A, Engelhardt B, D'Apolito K, Bogen D, Lester B. Comparison of Safety and Efficacy of Methadone vs Morphine for Treatment of Neonatal Abstinence Syndrome: A Randomized Clinical Trial. JAMA Pediatr. 2018 Aug 1;172(8):741-748. doi: 10.1001/jamapediatrics.2018.1307. PMID 29913015
- [Background] Kraft WK, Adeniyi-Jones SC, Ehrlich ME. Buprenorphine for the Neonatal Abstinence Syndrome. N Engl J Med. 2017 Sep 7;377(10):997-998. doi: 10.1056/NEJMc1709121. No abstract available. PMID 28877016
- [Background] Brown MS, Hayes MJ, Thornton LM. Methadone versus morphine for treatment of neonatal abstinence syndrome: a prospective randomized clinical trial. J Perinatol. 2015 Apr;35(4):278-83. doi: 10.1038/jp.2014.194. Epub 2014 Oct 30. PMID 25357093
- [Background] Asti L, Magers JS, Keels E, Wispe J, McClead RE Jr. A quality improvement project to reduce length of stay for neonatal abstinence syndrome. Pediatrics. 2015 Jun;135(6):e1494-500. doi: 10.1542/peds.2014-1269. Epub 2015 May 4. PMID 25941308
- [Background] Devlin LA, Lau T, Radmacher PG. Decreasing Total Medication Exposure and Length of Stay While Completing Withdrawal for Neonatal Abstinence Syndrome during the Neonatal Hospital Stay. Front Pediatr. 2017 Oct 10;5:216. doi: 10.3389/fped.2017.00216. eCollection 2017. PMID 29067285
- [Background] Kraft WK, Dysart K, Greenspan JS, Gibson E, Kaltenbach K, Ehrlich ME. Revised dose schema of sublingual buprenorphine in the treatment of the neonatal opioid abstinence syndrome. Addiction. 2011 Mar;106(3):574-80. doi: 10.1111/j.1360-0443.2010.03170.x. Epub 2010 Oct 6. PMID 20925688
- [Background] Hall ES, Rice WR, Folger AT, Wexelblatt SL. Comparison of Neonatal Abstinence Syndrome Treatment with Sublingual Buprenorphine versus Conventional Opioids. Am J Perinatol. 2018 Mar;35(4):405-412. doi: 10.1055/s-0037-1608634. Epub 2017 Nov 7. PMID 29112997
- [Background] Moore JN, Gastonguay MR, Ng CM, Adeniyi-Jones SC, Moody DE, Fang WB, Ehrlich ME, Kraft WK. The Pharmacokinetics and Pharmacodynamics of Buprenorphine in Neonatal Abstinence Syndrome. Clin Pharmacol Ther. 2018 Jun;103(6):1029-1037. doi: 10.1002/cpt.1064. Epub 2018 Apr 28. PMID 29516490
- [Background] Anagnostis EA, Sadaka RE, Sailor LA, Moody DE, Dysart KC, Kraft WK. Formulation of buprenorphine for sublingual use in neonates. J Pediatr Pharmacol Ther. 2011 Oct;16(4):281-4. doi: 10.5863/1551-6776-16.4.281. PMID 22768012